CLINICAL TRIAL: NCT06606171
Title: Floor Sitting: an Exploration of Its Effects on Health and Sedentary Activity
Brief Title: Floor Sitting Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Pyatak (Other)
Responsible Party: Sponsor-Investigator, Beth Pyatak, Faculty Advisor, University of Southern California
Organization: University of Southern California (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: UP-24-00696
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Well-being/Quality of Life; Posture; Sedentary Behaviors
Keywords: sedentary behaviors; sitting behaviors; ergonomics; posture; floor sitting; accelerometry; movement
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Chair Sitting Experimental Arm (Experimental): Participants in this arm will undergo a 30-minute session of chair sitting in a non-swivel chair. Activities during this session include engaging in typical desk activities to simulate a natural office environment.
  Interventions: Behavioral: Chair Sitting (30 minutes)
- Floor Sitting Experimental Arm (Experimental): Participants in this arm will undergo a 30-minute session of floor sitting on a cushioned mat. They will engage in the same desk activities as the chair sitting arm to maintain consistency across conditions.
  Interventions: Behavioral: Floor Sitting (30 minutes)
- Extended Floor Sitting Intervention (Experimental): Participants in this arm will engage in daily floor sitting as part of their usual activities at home to assess the long-term effects of floor sitting on well-being and health.
  Interventions: Behavioral: Daily Floor Sitting Practice (1 month)

INTERVENTIONS:
Behavioral: Chair Sitting (30 minutes) — This intervention involves a single session of chair sitting for 30 minutes, where participants will sit in a standardized non-swivel chair and perform desk-based activities like computer use.
  Arms: Chair Sitting Experimental Arm
Behavioral: Floor Sitting (30 minutes) — This intervention entails a single session of floor sitting for 30 minutes, with participants seated on a cushioned mat performing similar desk activities as in the chair sitting session.
  Arms: Floor Sitting Experimental Arm
Behavioral: Daily Floor Sitting Practice (1 month) — Participants will be instructed to incorporate at least one hour of floor sitting into their daily routine for a duration of one month.
  Arms: Extended Floor Sitting Intervention

SUMMARY:
The goal of this clinical trial is to evaluate the impact of different sitting environments on general well-being and movement patterns in healthy young adults aged 18-35. The main questions it aims to answer are:

Does floor sitting lead to increased movement and postural changes compared to chair sitting? Over a month-long period, how does sustained floor sitting influence overall well-being, posture, and movement habits?

Researchers will compare the effects of chair sitting and floor sitting in a controlled lab environment (Aim 1) and observe the longer-term effects of habitual floor sitting in participants natural environments (Aim 2) to see if consistent floor sitting promotes more dynamic movement and comfort.

Participants will:

Undergo two 30-minute experimental sitting sessions, one in a chair and the other on the floor, while engaging in typical desk activities (Aim 1).

Participate in a month-long study where they integrate an hour of floor sitting into their daily routines, recording their experiences and any changes in sitting habits through daily diaries and in-depth interview (Aim 2).

ELIGIBILITY:
Inclusion Criteria:

* age 18-35 years
* English-speaking
* willing and able to complete study procedures.

Exclusion Criteria:

* Any injuries or conditions that would limit participants from sitting on the floor in a safe manner, mental states that would preclude the complete understanding of the protocol and compliance, and prior knowledge of the study hypotheses, as it may potentially influence participant behavior and compromise the integrity of the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Movement Patterns via Accelerometry | Recorded continuously during each 30-minute sitting session; analysis will compare aggregate data from the two sessions.
  Measurement of movement patterns using accelerometry to assess changes in physical activity levels and subtle movements, including frequency, intensity, and duration of movements during different sitting interventions (chair vs. floor sitting).
Variations in Sitting Posture Captured by Video Analysis | Postural data will be collected throughout the two 30-minute experimental sitting sessions, with comparative analysis conducted post-intervention.
  Utilization of video recordings to analyze and quantify postural changes during sitting sessions. This will involve evaluating variations in posture, such as shifts from upright to slouched positions, and identifying the frequency and diversity of postural transitions during each session.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Pyatak, Study Chair — University of Southern California
Locations (1):
- Lifestyle Redesign for Chronic Conditions Lab, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided